CLINICAL TRIAL: NCT05083338
Title: Prospective Evaluation of Psychological, Psychophysical and Epigenetic Determinants of Chronic Pain After Cytoreductive - Hyperthermic Intraoperative Chemotherapy in Adult Patients
Brief Title: Psychological, Psychophysical and Epigenetic Determinants of Chronic Pain After Cytoreductive - Hyperthermic Intraoperative Chemotherapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0027; NCI-2021-09684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0027 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Appendix Carcinoma; Carcinomatosis; Colorectal Carcinoma; Gastric Carcinoma; Malignant Peritoneal Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Appendiceal Neoplasms; Carcinoma; Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire, pain assessment, biospecimen): Patients complete questionnaires over 15 minutes and undergo pain assessments prior to surgery and at 3, 6 and 12 months after surgery. Patients also undergo blood sample collection before surgery and optionally at 3, 6 and 12 months after surgery.
  Interventions: Procedure: Biospecimen Collection; Procedure: Pain Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Pain Assessment — Undergo pain assessment
  Other Names: Pain Measurement
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study learns if depression, anxiety, and catastrophizing (thought patterns that prompt people to expect the worst) are associated with chronic pain after surgery among patients who are scheduled to have cytoreductive surgery with intraoperative hyperthermic chemotherapy. Information from this study may improve the understanding of persistent and chronic postsurgical pain integrating multiple layers of biological and behavioral sciences.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the association of preoperative psychological risk factors (depression, anxiety or catastrophizing) with the development of chronic postsurgical pain after cytoreductive surgery with intraoperative hyperthermic chemotherapy (CRS-HIPEC).

SECONDARY OBJECTIVES:

I. To evaluate the association of preoperative psychological risk factors (depression, anxiety or catastrophizing) with the development of persistent postsurgical pain after CRS-HIPEC.

II. To evaluate the association between preoperative abnormal sensory disturbances and chronic postsurgical pain after CRS-HIPEC.

III. To assess the association of blood micro ribonucleic acids (RNAs) signatures with the development of chronic postsurgical pain after CRS-HIPEC.

IV. To determine the rate of and factors associated with persistent and chronic opioid use after CRS-HIPEC.

V. To determine the rate of persistent and chronic postsurgical anxiety and depression.

VI. To investigate changes in psychological risk factors (depression, anxiety or catastrophizing) and sensory disturbances after CRS-HIPEC overtime.

EXPLORATORY OBJECTIVE:

I. To explore the impact of perioperative (in-patient) opioid use, non-opioid analgesic use and anesthetics on the development of persistent and chronic opioid use after CRS-HIPEC.

OUTLINE:

Patients complete questionnaires over 15 minutes and undergo pain assessments prior to surgery and at 3, 6 and 12 months after surgery. Patients also undergo blood sample collection before surgery and optionally at 3, 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; with or without history of preoperative abdominal pain
* American Society of Anesthesiologists physical status (ASA) 1-4
* Scheduled surgery: open CRS-HIPEC surgery for primary peritoneal malignancy or secondary carcinomatosis (i.e., appendiceal, colorectal and gastric cancers)
* Written informed consent

Exclusion Criteria:

* ASA >= 4 or emergency surgeries
* Patients with extra-abdominal metastatic disease
* Patients cognitive or neurologically unable to complete questionnaires preoperatively
* Non-English-speaking patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without history of preoperative abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Chronic postsurgical pain | through study completion, an average of 1 year
  Defined as pain that develops or increases in intensity compared to preoperative after cyotreductive surgery with intraoperative hyperthermic chemotherapy (CRS-HIPEC), lasts for more than 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Cata, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org